CLINICAL TRIAL: NCT03951077
Title: Phase 2, Multicenter, Double-blind (Sponsor-unblinded), Randomized, Placebo-Controlled Study of the Safety and Efficacy of Elagolix in Women With Polycystic Ovary Syndrome
Brief Title: Study of the Safety and Efficacy of Elagolix in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M16-837
Record Dates: First submitted 2019-05-06; First posted 2019-05-15 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Hormone; Elagolix
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Placebo (Placebo Comparator): Placebo taken orally twice a day (BID)
  Interventions: Drug: Placebo
- Elagolix 25 mg BID (Experimental): Elagolix 25 mg taken orally BID plus placebo
  Interventions: Drug: Elagolix; Drug: Placebo
- Elagolix 50 mg Once Daily (QD) (Experimental): Elagolix 50 mg taken orally QD plus placebo
  Interventions: Drug: Elagolix; Drug: Placebo
- Elagolix 75 mg BID (Experimental): Elagolix 75 mg taken orally BID plus placebo
  Interventions: Drug: Elagolix; Drug: Placebo
- Elagolix 150 mg QD (Experimental): Elagolix 150 mg taken orally QD plus placebo
  Interventions: Drug: Elagolix; Drug: Placebo
- Elagolix 300 mg QD (Experimental): Elagolix 300 mg taken orally QD plus placebo
  Interventions: Drug: Elagolix; Drug: Placebo

INTERVENTIONS:
Drug: Elagolix — Capsule administered orally
  Other Names: Orilissa
  Arms: Elagolix 150 mg QD; Elagolix 25 mg BID; Elagolix 300 mg QD; Elagolix 50 mg Once Daily (QD); Elagolix 75 mg BID
Drug: Placebo — Capsule administered orally

SUMMARY:
This study will assess the potential impact of elagolix on disordered pituitary and ovarian hormones in women with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
This is a phase 2, multicenter, double-blind (sponsor-unblinded), randomized, placebo-controlled study to assess the safety and efficacy of elagolix in women with PCOS. PCOS is one of the most common hormonal disorders in women of reproductive age, yet few treatment options are available. This study will help determine if elagolix can impact disordered hormonal dynamics in women with PCOS and at what dosage.

ELIGIBILITY:
Inclusion Criteria:

* Participants with clinical diagnosis of PCOS.
* Participants with a body mass index (BMI) of 18.5 to 38 kg/m^2 at time of Screening.

Exclusion Criteria:

* Participants with newly diagnosed medical condition requiring intervention that has not been stabilized at least 30 days prior to Baseline.
* Participants with a significant medical condition that require intervention during the course of study participation (such as anticipated major elective surgery).
* Participants with an unstable medical condition (including, but not limited to, uncontrolled hypertension, epilepsy requiring anti-epileptic medicine, unstable angina, confirmed inflammatory bowel disease, hyperprolactinemia, clinically significant infection or injury).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- United States (50):
  - Alabama Clinical Therapeutics /ID# 211498, Birmingham, Alabama
  - Mobile, OBGYN P.C. /ID# 205574, Mobile, Alabama
  - Medical Ctr for Clin Research /ID# 205694, San Diego, California
  - UCSF Center for Reproductive Health /ID# 210836, San Francisco, California
  - Avail Clinical Research /ID# 210873, DeLand, Florida
  - University of FL Southside Women's Specialists /ID# 210872, Jacksonville, Florida
  - Segal Institute for Clinical Research /ID# 205490, North Miami, Florida
  - A Premier Medical Research of FL /ID# 215659, Orange City, Florida
  - Virtus Research Consultant,LLC /ID# 205475, Wellington, Florida
  - Comprehensive Clinical Trials LLC /ID# 205458, West Palm Beach, Florida
  - Mount Vernon Clinical Res, LLC /ID# 205695, Atlanta, Georgia
  - Bingham Memorial Hospital /ID# 205606, Blackfoot, Idaho
  - Leavitt Womens Healthcare /ID# 205571, Idaho Falls, Idaho
  - Womens Healthcare Assoc, DBA /ID# 211528, Idaho Falls, Idaho
  - Sonora Clinical Research /ID# 205623, Meridian, Idaho
  - Asr, Llc /Id# 207037, Nampa, Idaho
  - PRN Professional Research Network of Kansas, LLC /ID# 205875, Wichita, Kansas
  - Clinical Trials Management, LLC - Covington /ID# 211219, Covington, Louisiana
  - Clinical Trials Management, LLC - Metairie /ID# 205494, Metairie, Louisiana
  - Baltimore Suburban Health /ID# 205619, Baltimore, Maryland
  - Johns Hopkins University /ID# 205617, Baltimore, Maryland
  - Capital Women's Care - Frederi /ID# 210276, Frederick, Maryland
  - NECCR Fall River LLC /ID# 205567, Fall River, Massachusetts
  - Wayne State University Physician Group - Southfield /ID# 210245, Southfield, Michigan
  - Private practice: Dr. Rex G. Mabey JR /ID# 211149, Las Vegas, Nevada
  - Dr. Nader and Associates M.D. P.C. /ID# 211150, North Las Vegas, Nevada
  - Cooper University Hospital/Sheridan Pavilion /ID# 205576, Marlton, New Jersey
  - University of New Mexico /ID# 212594, Albuquerque, New Mexico
  - SUNY Downstate Medical Center /ID# 211180, Brooklyn, New York
  - University of Rochester - Strong Fertility Center - Rochester /ID# 210328, Rochester, New York
  - OB.GYN Associates of WNY /ID# 210765, West Seneca, New York
  - Upstate Clinical Research Associates /ID# 205717, Williamsville, New York
  - Carolina Institute for Clinical Research - Fayetteville /ID# 211319, Fayetteville, North Carolina
  - Wake Forest Baptist Medical Center /ID# 211473, Winston-Salem, North Carolina
  - Duplicate_Aventiv Research, Inc. /ID# 205460, Columbus, Ohio
  - Univ Hosp Landerbrook /ID# 205558, Mayfield Heights, Ohio
  - AC Clinical Research /ID# 205492, Tiffin, Ohio
  - Penn State University and Milton S. Hershey Medical Center /ID# 205555, Hershey, Pennsylvania
  - Thomas Jefferson University /ID# 205614, Philadelphia, Pennsylvania
  - Reading Hospital /ID# 211322, Reading, Pennsylvania
  - Chattanooga Medical Research /ID# 215190, Chattanooga, Tennessee
  - WR-Medical Research Center of Memphis LLC /ID# 205636, Memphis, Tennessee
  - The University of Texas Southwestern Medical Center /ID# 210804, Dallas, Texas
  - University of Texas (UT) Health Women's Research Center at Memorial City /ID# 216266, Houston, Texas
  - Advances in Health, Inc. /ID# 211249, Houston, Texas
  - Duplicate_Diagnostic Clinic of Longview /ID# 211019, Longview, Texas
  - Center of Reproductive Medicine /ID# 211250, Webster, Texas
  - Virginia Mason - Seattle Orthapedics /ID# 205586, Seattle, Washington
  - Seattle Women's Health, Research, Gynecology /ID# 205569, Seattle, Washington
  - North Spokane Women's Health /ID# 205585, Spokane, Washington
- Puerto Rico (4):
  - Puerto Rico Medical Research /ID# 211104, Ponce
  - University of Puerto Rico, Medical Sciences Campus /ID# 212320, Rio Piedras
  - Duplicate_Rodriguez-Ginorio, San Juan /ID# 211105, San Juan
  - Mindful Medical Research /ID# 212323, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Snabes MC, Ng J, Li H, Ali I, Shebley M, Schlaff WD. Phase 2, double-blind, randomized, placebo-controlled study of the safety and efficacy of elagolix in women with polycystic ovary syndrome. F S Rep. 2023 Feb 21;4(2):206-212. doi: 10.1016/j.xfre.2023.02.007. eCollection 2023 Jun. PMID 37398623
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized 2:2:2:2:2:3 to the following treatments: 25 mg twice daily (BID), 50 mg once daily (QD), 75 mg BID, 150 mg QD, 300 mg QD, or placebo.
Groups:
- Placebo: Placebo taken orally BID
- Elagolix 50 mg QD: Elagolix 50 mg taken orally QD plus placebo
Period: Overall Study
Arm/Group | Placebo | Elagolix 25 mg BID | Elagolix 50 mg QD | Elagolix 75 mg BID | Elagolix 150 mg QD | Elagolix 300 mg QD
Started (Randomized) | 27 | 18 | 18 | 18 | 19 | 18
Randomized and Treated | 26 | 18 | 17 | 17 | 18 | 18
Completed | 9 | 4 | 5 | 6 | 3 | 7
Not Completed | 18 | 14 | 13 | 12 | 16 | 11
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0 | 3 | 3 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2 | 3 | 2 | 3
Not completed — Non-Compliance With Study Procedures | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other, Not Specified | 12 | 10 | 10 | 5 | 9 | 6
Not completed — Did Not Receive Any Study Drug | 1 | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix 25 mg BID | Elagolix 50 mg QD | Elagolix 75 mg BID | Elagolix 150 mg QD | Elagolix 300 mg QD | Total
Number analyzed (Participants) | 26 | 18 | 17 | 17 | 18 | 18 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (4.60) | 25.3 (5.19) | 27.6 (4.85) | 26.9 (3.27) | 25.1 (4.19) | 26.1 (4.35) | 26.5 (4.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 17 | 17 | 18 | 18 | 114
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 6 | 3 | 4 | 4 | 27
  Not Hispanic or Latino | 21 | 13 | 11 | 14 | 14 | 14 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 6 | 4 | 1 | 5 | 7 | 4 | 27
  White | 19 | 13 | 16 | 12 | 11 | 14 | 85
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  < 30 kg/m^2 | 8 | 5 | 5 | 5 | 5 | 5 | 33
  ≥ 30 kg/m^2 | 18 | 13 | 12 | 12 | 13 | 13 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Menstrual Cycle Responders
Description: A participant was considered a menstrual cycle responder if she has at least 2 normal menstrual cycles during the final 4 months of the treatment period. In addition, a participant was considered a complete menstrual cycle responder if she has normal menstrual cycles beginning at or before Month 3 that are maintained through Month 6 during the treatment period.
Time Frame: Week 0 (Baseline) to Week 24 (Month 6)
Population: Full Analysis Set: all randomly assigned participants who have received at least one dose of study drug in this study. Based on observed cases only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 25 mg BID | Elagolix 50 mg QD | Elagolix 75 mg BID | Elagolix 150 mg QD | Elagolix 300 mg QD
Number analyzed (Participants) | 26 | 18 | 17 | 17 | 18 | 18
percentage of participants | 7.7 [0.00 to 16.29] | 0 [0.00 to 0.00] | 0 [0.00 to 0.00] | 0 [0.00 to 0.00] | 0 [0.00 to 0.00] | 5.6 [0.00 to 14.44]
Statistical Analysis 1: Comparison: Placebo vs Elagolix 25 mg BID; Across the strata, 90% confidence interval (CI) for adjusted difference and p-value were calculated according to the Cochran-Mantel-Haenszel (CMH) test adjusted for strata (Baseline FG score [< 8, ≥ 8], and baseline normal/obese status [BMI < 30, ≥ 30]) for the comparison of between each elagolix group and placebo. If zero frequency occurred, the zero count was replaced by 0.1 to prevent dividing by zero; Test type: Superiority; p = 0.300, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = -5.9, 90% CI 2-sided [-15.38 to 3.49]
Statistical Analysis 2: Comparison: Placebo vs Elagolix 50 mg QD; Across the strata, 90% CI for adjusted difference and p-value were calculated according to the CMH test adjusted for strata (Baseline FG score [< 8, ≥ 8], and baseline normal/obese status [BMI < 30, ≥ 30]) for the comparison of between each elagolix group and placebo. If zero frequency occurred, the zero count was replaced by 0.1 to prevent dividing by zero; Test type: Superiority; p = 0.320, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = -5.9, 90% CI 2-sided [-15.65 to 3.86]
Statistical Analysis 3: Comparison: Placebo vs Elagolix 75 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.315, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = -5.6, 90% CI 2-sided [-14.87 to 3.59]
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.265, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = -6.7, 90% CI 2-sided [-16.63 to 3.19]
Statistical Analysis 5: Comparison: Placebo vs Elagolix 300 mg QD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.914, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = -0.8, 90% CI 2-sided [-13.10 to 11.48]

2. Secondary Outcome: Change From Baseline in Area Under the Luteinizing Hormone (LH) Serum Concentration-time Curve (AUC) at Week 1
Time Frame: Week 0 (Baseline), Week 1: before the morning dose (0 hour) and at 0.5 (± 5 minutes), 1 (± 5 minutes), 1.5 (± 5 minutes), 2 (± 15 minutes), 2.5 (± 15 minutes), 3 (± 15 minutes), 3.5 (± 15 minutes), and 4 (± 15 minutes) hours after dosing.
Population: Full Analysis Set: all randomly assigned participants who have received at least one dose of study drug in this study. Participants with an assessment.
Measure: Least Squares Mean (Standard Error); unit: (IU/L)*hr
Arm/Group | Placebo | Elagolix 25 mg BID | Elagolix 50 mg QD | Elagolix 75 mg BID | Elagolix 150 mg QD | Elagolix 300 mg QD
Number analyzed (Participants) | 24 | 15 | 15 | 16 | 13 | 15
(IU/L)*hr | -1.82 (2.292) | -7.75 (2.867) | -10.65 (2.861) | -17.92 (2.692) | -7.97 (3.112) | -13.54 (2.763)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 25 mg BID; P-value is from mixed-effect model repeated measure (MMRM) with the fixed categorical effects of treatment, visit, treatment-by-visit interaction, baseline FG score (< 8, ≥ 8), and baseline normal/obese status (BMI < 30, ≥ 30), participant as a random effect, and the continuous fixed covariate of baseline measurement. Model is based on unstructured variance covariance structure; Test type: Superiority; p = 0.087, MMRM; Least Squares (LS) Mean of Difference = -5.93, 90% CI 2-sided [-11.628 to -0.231], Standard Error of Mean 3.429
Statistical Analysis 2: Comparison: Placebo vs Elagolix 50 mg QD; P-value is from MMRM with the fixed categorical effects of treatment, visit, treatment-by-visit interaction, baseline FG score (< 8, ≥ 8), and baseline normal/obese status (BMI < 30, ≥ 30), participant as a random effect, and the continuous fixed covariate of baseline measurement. Model is based on unstructured variance covariance structure; Test type: Superiority; p = 0.012, MMRM; LS Mean of Difference = -8.83, 90% CI 2-sided [-14.533 to -3.118], Standard Error of Mean 3.435
Statistical Analysis 3: Comparison: Placebo vs Elagolix 75 mg BID; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM; LS Mean of Difference = -16.10, 90% CI 2-sided [-21.673 to -10.519], Standard Error of Mean 3.356
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg QD; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.091, MMRM; LS Mean of Difference = -6.15, 90% CI 2-sided [-12.116 to -0.176], Standard Error of Mean 3.593
Statistical Analysis 5: Comparison: Placebo vs Elagolix 300 mg QD; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM; LS Mean of Difference = -11.72, 90% CI 2-sided [-17.418 to -6.016], Standard Error of Mean 3.431

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of treatment plus 30 days. Overall mean duration of treatment was 105.8 days.
Arm/Group | Placebo | Elagolix 25 mg BID | Elagolix 50 mg QD | Elagolix 75 mg BID | Elagolix 150 mg QD | Elagolix 300 mg QD
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/18 | 0/17 | 0/17 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/18 | 0/17 | 0/17 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 10/26 | 9/18 | 8/17 | 6/17 | 11/18 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Elagolix 25 mg BID (N=18) | Elagolix 50 mg QD (N=17) | Elagolix 75 mg BID (N=17) | Elagolix 150 mg QD (N=18) | Elagolix 300 mg QD (N=18)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Elagolix 25 mg BID (N=18) | Elagolix 50 mg QD (N=17) | Elagolix 75 mg BID (N=17) | Elagolix 150 mg QD (N=18) | Elagolix 300 mg QD (N=18)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
HYPERANDROGENISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SALIVARY GLAND CYST (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PILONIDAL CYST (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SCHISTOSOMIASIS CUTANEOUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAIL AVULSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD INSULIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BONE DENSITY DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIPIDS INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATTENTION DEFICIT HYPERACTIVITY DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MOOD SWINGS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STRESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC DISCOMFORT (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PREMENSTRUAL SYNDROME (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT03951077/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03951077/SAP_001.pdf